CLINICAL TRIAL: NCT02470585
Title: A Phase 3 Placebo-Controlled Study of Carboplatin/Paclitaxel With or Without Concurrent and Continuation Maintenance Veliparib (PARP Inhibitor) in Subjects With Previously Untreated Stages III or IV High-Grade Serous Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: Veliparib With Carboplatin and Paclitaxel and as Continuation Maintenance Therapy in Adults With Newly Diagnosed Stage III or IV, High-grade Serous, Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Acronym: VELIA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision not related to patient safety
Sponsor: AbbVie (Industry)
Collaborators: Australia New Zealand Gynaecological Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M13-694; 2014-005070-11 (EudraCT Number)
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Results first posted 2020-09-14 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Ovarian Cancer; Ovarian Neoplasm
Keywords: Veliparib; Carboplatin; Paclitaxel; Overall Survival; ABT-888; Randomized; Poly Adenosine Diphosphate (ADP) - Ribose Polymerase (PARP); Ovarian; BRCA; VELIA
MeSH Terms: conditions — Ovarian Neoplasms | interventions — veliparib; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | US Export: No

ARMS (3):
- Placebo + Carboplatin + Paclitaxel -> Placebo (Active Comparator): Participants will receive placebo to veliparib orally twice a day in combination with carboplatin/paclitaxel for six 21-day cycles followed by placebo monotherapy continuous dosing for an additional thirty 21-day cycles.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Other: Placebo to Veliparib
- Veliparib + Carboplatin + Paclitaxel -> Placebo (Experimental): Participants will receive 150 mg veliparib orally twice a day in combination with carboplatin/paclitaxel for six 21-day cycles followed by placebo monotherapy continuous dosing for an additional thirty 21-day cycles.
  Interventions: Drug: Veliparib; Drug: Paclitaxel; Drug: Carboplatin; Other: Placebo to Veliparib
- Veliparib + Carboplatin + Paclitaxel -> Veliparib (Experimental): Participants will receive 150 mg veliparib orally twice a day in combination with carboplatin/paclitaxel for six 21-day cycles followed by 300/400 mg veliparib monotherapy orally twice a day for an additional thirty 21-day cycles.
  Interventions: Drug: Veliparib; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Veliparib — Capsules for oral administration
  Other Names: ABT-888
  Arms: Veliparib + Carboplatin + Paclitaxel -> Placebo; Veliparib + Carboplatin + Paclitaxel -> Veliparib
Drug: Paclitaxel — Administered by intravenous infusion, either 80 mg/m² of body-surface area (BSA) on Days 1, 8, and 15 of each 21-day cycle (weekly dosing), or 175 mg/m² of BSA on Day 1 of each 21-day cycle (3-week dosing).
Drug: Carboplatin — Administered by intravenous infusion at an area under the curve (AUC) of 6 mg/mL/min every 3 weeks.
Other: Placebo to Veliparib — Capsules for oral administration
  Arms: Placebo + Carboplatin + Paclitaxel -> Placebo; Veliparib + Carboplatin + Paclitaxel -> Placebo

SUMMARY:
The primary objective of the study was to evaluate whether progression-free survival (PFS) was prolonged with the addition of veliparib to standard platinum-based chemotherapy (carboplatin/paclitaxel [C/P]) and continued as maintenance therapy compared with chemotherapy alone.

DETAILED DESCRIPTION:
Participants were randomized in a 1:1:1 ratio to one of three arms. Randomization in the entire population was stratified according to the timing of surgery and residual disease status (any residual disease after primary surgery vs. no residual disease after primary surgery vs. interval surgery) and the paclitaxel schedule (weekly vs. every 3 -weeks), stage of disease (III vs. IV), geographic region (Japan vs. North America and rest of world [ROW]), and germline breast cancer susceptibility gene (BRCA) mutation status (positive versus negative or Unknown).

Cytoreductive surgery could be performed before randomization and the initiation of study treatment (primary) or after 3 cycles of study treatment (interval). The weekly or every-3-week paclitaxel schedule and the choice of primary or interval cytoreductive surgery were determined at the discretion of the investigator.

The primary objective was evaluated in the BRCA-deficient cohort, participants with homologous recombination deficiency (HRD), and the intention-to-treat (ITT) population. These populations were sequentially inclusive, with the HRD population including the BRCA-deficient population, and the ITT population including the HRD and BRCA-deficient populations. The BRCA-deficient population was defined as participants with either a germline (gBRCA) and/or tissue-based (tBRCA) deleterious or suspected deleterious mutation in BRCA1 or BRCA2 confirmed by centralized testing. The HRD population was defined as participants with HRD tumors based on HRD score or presence of a deleterious or suspected deleterious mutation in BRCA1 or BRCA2 as determined by centralized testing.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of International Federation of Gynecology and Obstetrics (FIGO) Stage III or IV epithelial ovarian, fallopian tube, or primary peritoneal carcinoma, with the appropriate tissue available for histologic evaluation.
2. High-grade serous adenocarcinoma
3. Willing to undergo testing for gBRCA.
4. Adequate hematologic, renal, and hepatic function.
5. Neuropathy (sensory and motor) less than or equal to Grade 1.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
7. Participants who undergo primary cytoreductive surgery must be entered between 1 and 12 weeks after surgery. Participants undergoing interval surgery must have a tumor sample confirming the histological diagnosis prior to enrollment.
8. Participants with measurable disease or non-measurable disease are eligible. Participants may or may not have cancer-related symptoms.
9. Participant has one of the following available for pharmacodynamic analyses including somatic BRCA testing: Archived diagnostic formalin-fixed paraffin embedded (FFPE) tumor tissue; or tumor tissue biopsy collected prior to Cycle 1 Day 1.

Exclusion Criteria:

1. Endometrioid adenocarcinoma, carcinosarcoma, undifferentiated carcinoma, mixed epithelial adenocarcinoma, adenocarcinoma not otherwise specified, mucinous adenocarcinoma, clear cell adenocarcinoma, low-grade serous adenocarcinoma, or malignant Brenner's tumor.
2. Participants with synchronous primary endometrial cancer, or a past history of endometrial cancer unless all of the following conditions are met: endometrial cancer stage not greater than IA, no vascular or lymphatic invasion, no poorly differentiated subtypes including serous, clear cell, or other FIGO grade 3 lesions.
3. Participants with any evidence of other invasive malignancy being present within the last 3 years (with the exception of non-melanoma skin cancer). Participants are also excluded if their previous cancer treatment contraindicates this protocol's therapy.
4. Received prior radiotherapy to any portion of the abdominal cavity or pelvis.
5. Received prior chemotherapy for any abdominal or pelvic tumor.
6. Clinically significant uncontrolled condition(s).
7. Known history of allergic reaction to Cremophor-paclitaxel, carboplatin, Azo-Colourant Tartrazine (also known as FD&C Yellow 5 or E102), Azo-Colourant Orange Yellow-S (also known as FD&C Yellow 6 or E110) or known contraindications to any study supplied drug.
8. History or evidence upon physical examination of central nervous system (CNS) disease, including primary brain tumor, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) within 6 months of Cycle 1 Day 1.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1140 (Actual)
Dates: Start 2015-07-14 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2023-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (210):
- United States (135):
  - University of Alabama at Birmingham - Main /ID# 138087, Birmingham, Alabama
  - Tennessee Valley Gyn-Onc /ID# 139548, Huntsville, Alabama
  - University of South Alabama /ID# 138091, Mobile, Alabama
  - Alaska Womens Cancer Care /ID# 138231, Anchorage, Alaska
  - Arizona Oncology Associates, PC-HOPE /ID# 142002, Tucson, Arizona
  - Arizona Oncology Associates, PC-HOPE /ID# 143805, Tucson, Arizona
  - Arizona Oncology Associates, PC-HOPE /ID# 143806, Tucson, Arizona
  - Arizona Oncology Associates, PC-HOPE /ID# 143808, Tucson, Arizona
  - University of Arizona Cancer Center - North Campus /ID# 138084, Tucson, Arizona
  - University of Arizona Cancer Center - North Campus /ID# 139495, Tucson, Arizona
  - University of Arkansas for Medical Sciences /ID# 138253, Little Rock, Arkansas
  - John Muir Medical Center /ID# 139618, Concord, California
  - Ucsd /Id# 140323, La Jolla, California
  - Long Beach Memorial Medical Ct /ID# 147526, Long Beach, California
  - Kaiser Permanente /ID# 141305, Los Angeles, California
  - University of California, Los Angeles /ID# 138179, Los Angeles, California
  - Medical Oncology Care Assoc /ID# 139498, Orange, California
  - Univ CA, Irvine Med Ctr /ID# 139613, Orange, California
  - UC Davis Comprehensive Cancer Center - Main /ID# 144439, Sacramento, California
  - California Pacific Medical Ctr /ID# 138177, San Francisco, California
  - Kaiser Permanente - San Francisco /ID# 142051, San Francisco, California
  - Univ California, San Francisco /ID# 138178, San Francisco, California
  - Kaiser Permanente-Santa Clara /ID# 142053, Santa Clara, California
  - Stanford University School of Med /ID# 139450, Stanford, California
  - Palo Alto Medical Foundation /ID# 139452, Sunnyvale, California
  - Kaiser Permanente Medical Ctr-Vallejo /ID# 139492, Vallejo, California
  - Kaiser Permanente- Walnut Creek /ID# 142052, Walnut Creek, California
  - Kaiser Permanente, Waterpark III Institute for Health Research /ID# 139499, Aurora, Colorado
  - Univ of Colorado Cancer Center /ID# 138016, Aurora, Colorado
  - Hartford Healthcare /ID# 138184, New Britain, Connecticut
  - Yale University /ID# 138056, New Haven, Connecticut
  - University of Miami /ID# 139457, Miami, Florida
  - Sarasota Memorial Health Care /ID# 138180, Sarasota, Florida
  - Women's Cancer Associates /ID# 140321, St. Petersburg, Florida
  - Moffitt Cancer Center /ID# 138061, Tampa, Florida
  - Georgia Regents University /ID# 138085, Augusta, Georgia
  - IACT Health /ID# 138058, Columbus, Georgia
  - Memorial Health Univ Med Ctr /ID# 138019, Savannah, Georgia
  - St. Joseph's/Candler /ID# 138090, Savannah, Georgia
  - The Queens Medical Center /ID# 141709, Honolulu, Hawaii
  - Kapiolani Medical Center /ID# 140319, Honolulu, Hawaii
  - Rush University Medical Center /ID# 143491, Chicago, Illinois
  - University of Chicago /ID# 139612, Chicago, Illinois
  - NorthShore University HealthSystem - Evanston Hospital /ID# 139451, Evanston, Illinois
  - Sharma, Hinsdale, IL /ID# 140326, Hinsdale, Illinois
  - Advocate Lutheran General Hosp /ID# 139489, Park Ridge, Illinois
  - Indiana Univ School Medicine /ID# 139610, Indianapolis, Indiana
  - Saint Vincent /ID# 139537, Indianapolis, Indiana
  - McFarland Clinic, PC /ID# 139455, Ames, Iowa
  - University of Iowa Hospitals and Clinics /ID# 138082, Iowa City, Iowa
  - Univ Kansas Med Ctr /ID# 140322, Kansas City, Kansas
  - Baptist Health Lexington /ID# 139542, Lexington, Kentucky
  - University of Kentucky Chandler Medical Center /ID# 138060, Lexington, Kentucky
  - Norton Cancer Institute /ID# 139567, Louisville, Kentucky
  - MMP Women's Health /ID# 139544, Portland, Maine
  - Greater Baltimore Medical Ctr /ID# 138049, Baltimore, Maryland
  - Sinai Hospital of Baltimore /ID# 141306, Baltimore, Maryland
  - Weinberg Cancer Inst Franklin /ID# 138235, Rossville, Maryland
  - Baystate Medical Center /ID# 139456, Springfield, Massachusetts
  - UMass Memorial Medical Center /ID# 139458, Worcester, Massachusetts
  - Wayne State University /ID# 139601, Detroit, Michigan
  - Henry Ford Health System /ID# 139536, Detroit, Michigan
  - William Beaumont Hospital /ID# 139550, Royal Oak, Michigan
  - Mayo Clinic - Rochester /ID# 139565, Rochester, Minnesota
  - Mmcorc /Id# 139534, Saint Louis Park, Minnesota
  - St. Dominic Hospital /ID# 138241, Jackson, Mississippi
  - Ellis Fischel Cancer Center /ID# 139571, Columbia, Missouri
  - Cancer Research For the Ozarks /ID# 139538, Springfield, Missouri
  - Ferrell-Duncan Clinic /ID# 143484, Springfield, Missouri
  - Washington University-School of Medicine /ID# 138089, St Louis, Missouri
  - Nebraska Methodist Hospital /ID# 139600, Omaha, Nebraska
  - Womens Cancer Center of Nevada /ID# 138092, Las Vegas, Nevada
  - Renown Regional Medical Center /ID# 138237, Reno, Nevada
  - Dartmouth-Hitchcock Medical Center /ID# 139502, Lebanon, New Hampshire
  - MD Anderson Cancer Ctr at Coop /ID# 139616, Camden, New Jersey
  - Hackensack Univ Med Ctr /ID# 143776, Hackensack, New Jersey
  - University of New Mexico /ID# 144220, Albuquerque, New Mexico
  - SW Gynecologic Oncology Assoc /ID# 147097, Albuquerque, New Mexico
  - Women's Cancer Care Associates /ID# 138234, Albany, New York
  - SUNY Downstate Medical Center /ID# 139533, Brooklyn, New York
  - Roswell Park Comprehensive Cancer Center /ID# 138052, Buffalo, New York
  - Northwell Health /ID# 139572, Lake Success, New York
  - Icahn School of Med Mt. Sinai /ID# 139617, New York, New York
  - Columbia University Medical Center /ID# 138252, New York, New York
  - Memorial Sloan Kettering Cancer Center /ID# 138017, New York, New York
  - Memorial Sloan Kettering Cancer Center /ID# 154464, New York, New York
  - SUNY Upstate Medical University - Downtown /ID# 139513, Syracuse, New York
  - Montefiore Medical Center /ID# 139585, The Bronx, New York
  - Hope Womens Cancer Centers /ID# 139614, Asheville, North Carolina
  - Univ NC Chapel Hill /ID# 138547, Chapel Hill, North Carolina
  - Atrium Health Carolinas Medical Center /ID# 139568, Charlotte, North Carolina
  - Presbyterian Cancer Center /ID# 139590, Charlotte, North Carolina
  - Duke University Medical Center /ID# 138048, Durham, North Carolina
  - Wake Forest Baptist Medical Center /ID# 139588, Winston-Salem, North Carolina
  - University of Cincinnati /ID# 139619, Cincinnati, Ohio
  - Univ Hosp Cleveland /ID# 139615, Cleveland, Ohio
  - Fairview Hospital /ID# 144403, Cleveland, Ohio
  - Cleveland Clinic Main Campus /ID# 139501, Cleveland, Ohio
  - The Ohio State University - Columbus /ID# 138053, Columbus, Ohio
  - Columbus NCORP /ID# 139587, Columbus, Ohio
  - Womens Cancer Center /ID# 138062, Kettering, Ohio
  - Hillcrest Hospital /ID# 144404, Mayfield Heights, Ohio
  - Univ Oklahoma HSC /ID# 138020, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists /ID# 138059, Tulsa, Oklahoma
  - Willamette Valley Cancer Institute /ID# 140318, Eugene, Oregon
  - Kaiser Permanente, NW /ID# 138249, Portland, Oregon
  - Abington Memorial Hospital /ID# 138086, Abington, Pennsylvania
  - University of Pennsylvania /ID# 140079, Philadelphia, Pennsylvania
  - Thomas Jefferson University /ID# 138239, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center /ID# 149479, Philadelphia, Pennsylvania
  - University of Pittsburgh MC /ID# 138054, Pittsburgh, Pennsylvania
  - Reading Hospital /ID# 138057, Reading, Pennsylvania
  - Women and Infants Hospital /ID# 138083, Providence, Rhode Island
  - Medical University of South Carolina /ID# 138181, Charleston, South Carolina
  - Sanford Research/USD /ID# 139624, Sioux Falls, South Dakota
  - Chattanoogas Program in Womens /ID# 139545, Chattanooga, Tennessee
  - Texas Oncology - Austin Central /ID# 143817, Austin, Texas
  - Texas Oncology - South Austin /ID# 143818, Austin, Texas
  - Texas Oncology - Bedford /ID# 143814, Bedford, Texas
  - Texas Oncology - Medical City Dallas /ID# 143809, Dallas, Texas
  - Texas Oncology - Medical City Dallas /ID# 143812, Dallas, Texas
  - Texas Oncology - Forth Worth /ID# 143811, Fort Worth, Texas
  - Houston Methodist Hospital - Scurlock Tower /ID# 138232, Houston, Texas
  - Memorial Hermann Hospital /ID# 138238, Houston, Texas
  - Texas Oncology - The Woodlands /ID# 142003, The Woodlands, Texas
  - Texas Oncology - Tyler /ID# 143810, Tyler, Texas
  - University of Utah /ID# 138250, Salt Lake City, Utah
  - University of Vermont Medical Center /ID# 138251, Burlington, Vermont
  - University of Virginia /ID# 138088, Charlottesville, Virginia
  - Carilion Roanoke Memorial Hosp /ID# 139602, Roanoke, Virginia
  - Skagit Valley Medical Center /ID# 139586, Mount Vernon, Washington
  - MultiCare Regional Cancer Ctr /ID# 149872, Puyallup, Washington
  - Multicare Institute for Research and Innovation /ID# 143485, Tacoma, Washington
  - HSHS St. Vincent Hospital /ID# 139453, Green Bay, Wisconsin
  - Froedtert & the Medical College of Wisconsin /ID# 139449, Milwaukee, Wisconsin
- Australia (19):
  - Coffs Harbour Health Campus /ID# 145132, Coffs Harbour, New South Wales
  - Gosford Hospital /ID# 145299, Gosford, New South Wales
  - St George Hospital /ID# 145138, Kogarah, New South Wales
  - Newcastle Private Hospital /ID# 145834, Lambton Heights, New South Wales
  - The Prince of Wales Hospital /ID# 145134, Randwick, New South Wales
  - Northern Cancer Institute /ID# 145681, St Leonards, New South Wales
  - Calvary Mater Newcastle /ID# 145139, Waratah, New South Wales
  - Westmead Hospital /ID# 145137, Westmead, New South Wales
  - Southern Medical Day Care Ctr /ID# 145133, Wollongong, New South Wales
  - The Townsville Hospital /ID# 149163, Douglas, Queensland
  - Royal Brisbane and Women's Hospital /ID# 145135, Herston, Queensland
  - Icon Cancer Centre /ID# 148208, South Brisbane, Queensland
  - Mater Misericordiae Limited /ID# 145682, South Brisbane, Queensland
  - Royal Adelaide Hospital /ID# 150071, Adelaide, South Australia
  - Monash Health /ID# 145297, Clayton, Victoria
  - Cabrini Health /ID# 145142, Malvern, Victoria
  - Royal Womens Hospital /ID# 145136, Parkville, Victoria
  - Sir Charles Gairdner Hospital /ID# 145140, Nedlands, Western Australia
  - St. John of God Subiaco Hosp /ID# 147742, Subiaco, Western Australia
- Brazil (5):
  - Hc Ufmg /Id# 137156, Belo Horizonte, Minas Gerais
  - Hospital Sao Lucas da PUCRS /ID# 137157, Porto Alegre, Rio Grande do Sul
  - Hospital de Cancer de Barretos /ID# 137121, Barretos, São Paulo
  - Centro de Referencia da Saude da Mulher - Hospital Perola Byington /ID# 137120, São Paulo, São Paulo
  - Instituto Nacional de Câncer José de Alencar Gomes da Silva (INCA) /ID# 137155, Rio de Janeiro
- Denmark (2):
  - Vejle Sygehus /ID# 137262, Vejle, Region Syddanmark
  - Regionshospitalet Herning /ID# 137260, Herning
- Israel (6):
  - Rambam Health Care Campus /ID# 137434, Haifa
  - The Lady Davis Carmel MC /ID# 137537, Haifa
  - Shaare Zedek Medical Center /ID# 137435, Jerusalem
  - Meir Medical Center /ID# 139397, Kfar Saba
  - Sheba Medical Center /ID# 137436, Ramat Gan
  - Kaplan Medical Center /ID# 137536, Rehovot
- Japan (22):
  - Aichi Cancer Center Hospital /ID# 148398, Nagoya, Aichi-ken
  - National Hospital Organization Kyushu Cancer Center /ID# 149133, Fukuoka, Fukuoka
  - Kurume University Hospital /ID# 148697, Kurume-shi, Fukuoka
  - Iwate Medical University Hospital /ID# 147721, Shiwa-gun, Iwate
  - Kumamoto University Hospital /ID# 154169, Kumamoto, Kumamoto
  - Mie University Hospital /ID# 149169, Tsu, Mie-ken
  - Tohoku University Hospital /ID# 149818, Sendai, Miyagi
  - Niigata University Medical & Dental Hospital /ID# 149488, Niigata, Niigata
  - Kindai University Hospital /ID# 154947, Ōsaka-sayama, Osaka
  - Shizuoka Cancer Center /ID# 147723, Sunto-gun, Shizuoka
  - The Cancer Institute Hosp JFCR /ID# 148436, Koto-ku, Tokyo
  - Keio University Hospital /ID# 148326, Shinjuku-ku, Tokyo
  - Yamagata University Hospital /ID# 153646, Yamagata, Yamagata
  - Hyogo Cancer Center /ID# 148327, Akashi
  - Kansai Rosai Hospital /ID# 149237, Amagasaki
  - The Jikei Univ. Kashiwa Hosp. /ID# 149238, Kashiwa-shi
  - St. Marianna Univ Hospital /ID# 149327, Kawasaki
  - NHO Kure Medical Center and Ch /ID# 148569, Kure
  - Shikoku Cancer Center /ID# 148382, Matsuyama
  - Osaka International Cancer Institute /ID# 150778, Osaka
  - Hokkaido Cancer Center /ID# 148570, Sapporo
  - The Jikei University Hospital /ID# 148691, Tokyo
- Auckland City Hospital /ID# 145123, Auckland, New Zealand
- Uniwersyteckie C. Kliniczne /ID# 138021, Gdansk, Poland
- South Korea (6):
  - National Cancer Center /ID# 139404, Goyang, Gyeonggido
  - Korea University Anam Hospital /ID# 136908, 성북구, Gyeonggido
  - Gangnam Severance Hospital /ID# 136835, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 136834, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital /ID# 136909, Seoul
  - Asan Medical Center /ID# 136836, Seoul
- Spain (7):
  - Hospital Duran i Reynals /ID# 137298, L'Hospitalet de Llobregat, Barcelona
  - Hospital Univ Vall d'Hebron /ID# 137297, Barcelona
  - Hospital Clinic de Barcelona /ID# 137300, Barcelona
  - Hospital Clin Univ San Carlos /ID# 137402, Madrid
  - Hosp Univ 12 de Octubre /ID# 137299, Madrid
  - Hosp Univ Madrid Sanchinarro /ID# 137414, Madrid
  - Fundacion Inst Valenciano Onc /ID# 137403, Valencia
- United Kingdom (6):
  - Norfolk and Norwich Univ Hosp /ID# 137969, Norwich, Norfolk
  - Beatson west of scotland cancer center /ID# 137965, Glasgow, Scotland
  - Ninewells Hospital /ID# 137967, Dundee
  - James Paget University Hosp /ID# 137970, Great Yarmouth
  - Imanova Limited, Hammersmith Hospital /ID# 137966, London
  - Oxford Univ Hosp NHS Trust /ID# 137973, Oxford

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Background] Coleman RL, Fleming GF, Brady MF, Swisher EM, Steffensen KD, Friedlander M, Okamoto A, Moore KN, Efrat Ben-Baruch N, Werner TL, Cloven NG, Oaknin A, DiSilvestro PA, Morgan MA, Nam JH, Leath CA 3rd, Nicum S, Hagemann AR, Littell RD, Cella D, Baron-Hay S, Garcia-Donas J, Mizuno M, Bell-McGuinn K, Sullivan DM, Bach BA, Bhattacharya S, Ratajczak CK, Ansell PJ, Dinh MH, Aghajanian C, Bookman MA. Veliparib with First-Line Chemotherapy and as Maintenance Therapy in Ovarian Cancer. N Engl J Med. 2019 Dec 19;381(25):2403-2415. doi: 10.1056/NEJMoa1909707. Epub 2019 Sep 28. PMID 31562800
- [Derived] Swisher EM, Aghajanian C, O'Malley DM, Fleming GF, Kaufmann SH, Levine DA, Birrer MJ, Moore KN, Spirtos NM, Shahin MS, Reid TJ, Friedlander M, Steffensen KD, Okamoto A, Sehgal V, Ansell PJ, Dinh MH, Bookman MA, Coleman RL. Impact of homologous recombination status and responses with veliparib combined with first-line chemotherapy in ovarian cancer in the Phase 3 VELIA/GOG-3005 study. Gynecol Oncol. 2022 Feb;164(2):245-253. doi: 10.1016/j.ygyno.2021.12.003. Epub 2021 Dec 11. PMID 34906376
- [Derived] Washington CR, Moore KN. PARP inhibitors in the treatment of ovarian cancer: a review. Curr Opin Obstet Gynecol. 2021 Feb 1;33(1):1-6. doi: 10.1097/GCO.0000000000000675. PMID 33369580
- [Derived] Nishikawa T, Matsumoto K, Tamura K, Yoshida H, Imai Y, Miyasaka A, Onoe T, Yamaguchi S, Shimizu C, Yonemori K, Shimoi T, Yunokawa M, Xiong H, Nuthalapati S, Hashiba H, Kiriyama T, Leahy T, Komarnitsky P, Fujiwara K. Phase 1 dose-escalation study of single-agent veliparib in Japanese patients with advanced solid tumors. Cancer Sci. 2017 Sep;108(9):1834-1842. doi: 10.1111/cas.13307. Epub 2017 Aug 5. PMID 28665051

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at 188 sites in 10 countries (Australia, Brazil, Denmark, Israel, Japan, Poland, Republic of Korea, Spain, United Kingdom, and United States).
Pre-assignment Details: Participants were randomized in a 1:1:1 ratio to one of three treatment groups. Randomization was stratified according to the timing of surgery and residual disease after primary surgery or interval surgery, the paclitaxel schedule, stage of disease, geographic region, and germline breast cancer susceptibility gene (BRCA) mutation status.
Groups:
- Placebo + Carboplatin + Paclitaxel -> Placebo: Participants received placebo to veliparib orally twice a day in combination with carboplatin given at an area under the curve (AUC) of 6 milligrams per milliliter per minute (mg/mL/min) every 3 weeks, and paclitaxel 175 mg per square meter (mg/m²) of body-surface area (BSA), administered every 3 weeks, or 80 mg/m² administered weekly, for six 21-day cycles.
  Participants who completed chemotherapy without disease progression received matching placebo twice daily for an additional thirty 21-day cycles of maintenance therapy.
- Veliparib + Carboplatin + Paclitaxel -> Placebo: Participants received 150 mg veliparib orally twice a day in combination with carboplatin given at an AUC of 6 mg/mL/min every 3 weeks, and paclitaxel 175 mg/m² of BSA administered every 3 weeks, or 80 mg/m² administered weekly, for six 21-day cycles.
  Participants who completed chemotherapy without disease progression received matching placebo twice daily for an additional thirty 21-day cycles of maintenance therapy.
- Veliparib + Carboplatin + Paclitaxel -> Veliparib: Participants received 150 mg veliparib orally twice a day in combination with carboplatin given at an AUC of 6 mg/mL/min every 3 weeks, and paclitaxel 175 mg/m² of BSA administered every 3 weeks, or 80 mg/m² administered weekly, for six 21-day cycles.
  Participants who completed chemotherapy without disease progression received single-agent veliparib at a dose of 300 mg twice daily for 2 weeks (transition period) and then 400 mg veliparib twice daily if the dose in the transition period was not associated with limiting side effects for an additional thirty 21-day cycles of maintenance therapy.
Period: Overall Study
Arm/Group | Placebo + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Veliparib
Started | 375 | 383 | 382
Completed | 0 | 0 | 0
Not Completed | 375 | 383 | 382
Not completed — Death | 224 | 227 | 199
Not completed — Withdrew consent | 21 | 22 | 31
Not completed — Lost to Follow-up | 8 | 15 | 13
Not completed — Sponsor discontinued study | 117 | 110 | 122
Not completed — Other, not specified | 5 | 7 | 14
Not completed — Missing due to site non-compliance | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Population: The intention-to-treat (ITT) population consisted of all randomized participants.
Groups:
- Placebo + Carboplatin + Paclitaxel -> Placebo: Participants received placebo to veliparib orally twice a day in combination with carboplatin given at an area under the curve [AUC] of 6 mg per milliliter per minute (mg/mL/min), every 3 weeks, and paclitaxel 175 mg per square meter (mg/m²) of body-surface area (BSA), administered every 3 weeks, or 80 mg/m² administered weekly, for six 21-day cycles.
  Participants who completed chemotherapy without disease progression received matching placebo twice daily for an additional thirty 21-day cycles of maintenance therapy.
- Total: Total of all reporting groups
Arm/Group | Placebo + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Veliparib | Total
Number analyzed (Participants) | 375 | 383 | 382 | 1140
Age, Continuous [Median (Full Range); unit: years] | 62.0 [33.0 to 86.0] | 62.0 [22.0 to 88.0] | 62.0 [30.0 to 85.0] | 62.0 [22.0 to 88.0]
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 233 | 226 | 228 | 687
  ≥ 65 years | 142 | 157 | 154 | 453
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 375 | 383 | 382 | 1140
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 27 | 26 | 81
  Not Hispanic or Latino | 347 | 356 | 356 | 1059
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 299 | 297 | 300 | 896
  Black or African American | 10 | 13 | 20 | 43
  Asian | 59 | 69 | 56 | 184
  American Indian or Alaska Native | 1 | 1 | 1 | 3
  Native Hawaiian or other Pacific Islander | 1 | 0 | 2 | 3
  Multi-race | 3 | 0 | 0 | 3
  Missing | 2 | 3 | 3 | 8
Geographic Region [Count of Participants; unit: Participants]
  North America | 266 | 261 | 267 | 794
  Japan | 23 | 30 | 25 | 78
  Rest of World | 86 | 92 | 90 | 268
BRCA-Deficient Status [Count of Participants; unit: Participants] — The BRCA-mutation cohort was defined as participants who had deleterious or suspected deleterious germline (gBRCA) or tissue-based (tBRCA) mutations as determined by the Myriad BRACAnalysis® companion diagnostic (CDx) or myChoice® HRD CDx assay, respectively, in BRCA1 or BRCA2.
  Participants
    Germline or tissue BRCA1/2 mutation | 92 | 98 | 108 | 298
    Germline or tissue BRCA1/2 wildtype | 254 | 243 | 245 | 742
    Missing | 29 | 42 | 29 | 100
Homologous Recombination Deficiency (HRD) Status [Count of Participants; unit: Participants] — The HRD cohort consisted of participants who had tumors that were BRCA-mutated or had HRD according to the Myriad myChoice® assay, on which a score of ≥ 33 was considered to indicate HRD status, and a score of < 33 was considered to indicate non-HRD status.
  Participants
    HRD | 207 | 206 | 214 | 627
    Non-HRD | 124 | 123 | 125 | 372
    Missing | 44 | 54 | 43 | 141
Stage of Disease [Count of Participants; unit: Participants] — Staging of primary ovarian carcinomas according to the International Federation of Gynecology and Obstetrics (FIGO) criteria, based on clinical examination, surgical exploration, histologic characteristics and cytologic testing.
  STAGE III: Tumor involves 1 or both ovaries with cytologically or histologically confirmed spread to the peritoneum outside the pelvis and/or metastases to the retroperitoneal lymph nodes.
  STAGE IV: Distant metastases excluding peritoneal metastases
  Participants
    Stage III | 292 | 288 | 295 | 875
    Stage IV | 82 | 94 | 87 | 263
    Missing | 1 | 1 | 0 | 2
Type of Surgery Received [Count of Participants; unit: Participants] — Cytoreductive surgery could be performed before randomization and the initiation of study treatment (primary) or after 3 cycles of study treatment (interval), determined at the discretion of the investigator.
  Participants
    Primary | 250 | 253 | 261 | 764
    Interval | 107 | 114 | 99 | 320
    No surgery received | 18 | 16 | 22 | 56
Residual Disease After Primary Surgery [Count of Participants; unit: Participants] — Data were collected after interval surgery after cycle 3. Population: Participants who underwent primary surgery
  Participants
    number analyzed (Participants) | 250 | 253 | 261 | 764
    No residual disease | 116 | 118 | 124 | 358
    Microscopic residual disease only | 58 | 46 | 54 | 158
    Any macroscopic residual disease | 76 | 89 | 83 | 248
Residual Disease After Interval Surgery [Count of Participants; unit: Participants] — Population: Participants who underwent interval surgery
  Participants
    number analyzed (Participants) | 107 | 114 | 99 | 320
    No residual disease | 50 | 46 | 45 | 141
    Microscopic residual disease only | 22 | 30 | 24 | 76
    Any macroscopic residual disease | 31 | 34 | 27 | 92
    Missing | 4 | 4 | 3 | 11
Paclitaxel Dosing Regimen [Count of Participants; unit: Participants]
  Weekly | 193 | 203 | 190 | 586
  Every 3 weeks | 179 | 178 | 189 | 546
  Missing | 3 | 2 | 3 | 8
Germline BRCA Status [Count of Participants; unit: Participants]
  Germline BRCA1/2 mutation | 63 | 71 | 80 | 214
  Germline BRCA1/2 wildtype | 305 | 305 | 298 | 908
  Missing | 7 | 7 | 4 | 18

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) in the BRCA-deficient Population (Arm 3 vs Arm 1)
Description: PFS was defined as the time from the date that the participant was randomized to the date the participant experienced an event of disease progression, according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.1 (as determined by the investigator) or to the date of death if disease progression was not reached. If the participant did not have an event of disease progression or death prior to the analysis cut-off date, the participant's data were censored at the date of their last evaluable disease assessment. PFS was estimated using the Kaplan-Meier method. The analysis of PFS occurred when the protocol-specified number of PFS events was reached.
  Progressive Disease (PD): At least a 20% increase in the size of target lesions, compared with the smallest size recorded since the treatment started, and an absolute increase of ≥ 5 mm, or unequivocal progression of existing non-target lesions or the appearance of new lesions.
Time Frame: From randomization until the primary analysis data cut-off date of 03 May 2019, the median duration of follow-up was 28 months.
Population: Analyses were performed in 3 sequentially inclusive populations. The first analysis was conducted using the BRCA-mutation cohort which included participants with either a gBRCA and/or tBRCA deleterious or suspected deleterious mutation in BRCA1 or BRCA2.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Veliparib
Number analyzed (Participants) | 92 | 98 | 108
months | 22.0 [17.8 to 29.1] | 21.1 [17.0 to 25.5] | 34.7 [31.8 to NA] — Could not be estimated due to the low number of events
Statistical Analysis 1: Comparison: Placebo + Carboplatin + Paclitaxel -> Placebo vs Veliparib + Carboplatin + Paclitaxel -> Veliparib; The primary efficacy analyses compared investigator-assessed PFS in the Veliparib + Carboplatin + Paclitaxel -> Veliparib group (Arm 3) vs. the Placebo + Carboplatin + Paclitaxel -> Placebo group (Arm 1); Test type: Superiority — Multiplicity considerations included 3 treatment arms, (2 pairwise comparisons), 3 sequentially inclusive populations (BRCA-mutation population, HRD population, and ITT population), and multiple endpoints. A fixed-sequence testing procedure was used to control the Type I error rate at 0.05 from the primary efficacy endpoints sequentially through the secondary efficacy endpoints; p < 0.001, Log Rank — A 2-sided p-value of ≤ 0.05 was considered statistically significant in the following hierarchical testing sequence: PFS was to be compared first in the BRCA-mutation cohort, then in the HRD cohort, and then in the ITT population; Stratified according to residual disease status and disease stage; Hazard Ratio (HR) = 0.435, 95% CI 2-sided [0.277 to 0.683] — Cox proportional hazards model stratified according to the same factors as those used in the log-rank test above

2. Primary Outcome: Progression-Free Survival (PFS) in the Homologous Recombination Deficiency Cohort (Arm 3 vs Arm 1)
Description: PFS was defined as the time from the date that the participant was randomized to the date the participant experienced an event of disease progression, according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.1 (as determined by the investigator) or to the date of death if disease progression was not reached. If the participant did not have an event of disease progression or death, the participant's data were censored at the date of their last evaluable disease assessment. PFS was estimated using the Kaplan-Meier method. The primary analysis of PFS occurred when the protocol-specified number of PFS events was reached and was performed in 3 sequentially inclusive populations.
  Progressive Disease (PD): At least a 20% increase in the size of target lesions, compared with the smallest size recorded since the treatment started, and an absolute increase of ≥ 5 mm, or unequivocal progression of existing non-target lesions or the appearance of new lesions.
  .
Time Frame: as for outcome 1
Population: Analyses were performed in 3 sequentially inclusive populations. The second analysis was conducted using the HRD cohort which included participants in the BRCA-mutation cohort and those determined to have HRD tumors.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Veliparib
Number analyzed (Participants) | 207 | 206 | 214
months | 20.5 [17.8 to 22.8] | 18.1 [16.4 to 22.7] | 31.9 [25.8 to 38.0]
Statistical Analysis 1: Comparison: Placebo + Carboplatin + Paclitaxel -> Placebo vs Veliparib + Carboplatin + Paclitaxel -> Veliparib; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Log Rank — [p-value comment as in outcome 1, analysis 1]; Stratified according to residual disease status and disease stage; Hazard Ratio (HR) = 0.572, 95% CI 2-sided [0.433 to 0.756] — Cox proportional hazards model stratified according to the same factors as those used in the log-rank test above

3. Primary Outcome: Progression-Free Survival (PFS) in the Intention-to-treat Population (Arm 3 vs Arm 1)
Description: PFS was defined as the time from the date that the participant was randomized to the date the participant experienced an event of disease progression, according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.1 (as determined by the investigator) or to the date of death (all causes of mortality) if disease progression was not reached. If the participant did not have an event of disease progression according to RECIST criteria (as or death, the participant's data were censored at the date of their last evaluable disease assessment. PFS was estimated using the Kaplan-Meier method.
  Progressive Disease (PD): At least a 20% increase in the size of target lesions, compared with the smallest size recorded since the treatment started, and an absolute increase of ≥ 5 mm, or unequivocal progression of existing non-target lesions or the appearance of new lesions.
  The primary analysis of PFS occurred when the protocol-specified number of PFS events was reached.
Time Frame: as for outcome 1
Population: Analyses were performed in 3 sequentially inclusive populations. The third analysis was conducted using the intention-to-treat (ITT) population (all randomized participants).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Veliparib
Number analyzed (Participants) | 375 | 383 | 382
months | 17.3 [15.1 to 19.1] | 15.2 [14.1 to 17.3] | 23.5 [19.3 to 26.3]
Statistical Analysis 1: Comparison: Placebo + Carboplatin + Paclitaxel -> Placebo vs Veliparib + Carboplatin + Paclitaxel -> Veliparib; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Log Rank — [p-value comment as in outcome 1, analysis 1]; Stratified according to residual disease status and disease stage, choice of the paclitaxel regimen, and BRCA-mutation status; Hazard Ratio (HR) = 0.683, 95% CI 2-sided [0.562 to 0.831] — Cox proportional hazards model stratified according to the same factors as those used in the log-rank test above

4. Secondary Outcome: Progression-Free Survival (PFS) in the BRCA-deficient Population (Arm 2 vs Arm 1)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Veliparib
Number analyzed (Participants) | 92 | 98 | 108
months | 22.0 [17.8 to 29.1] | 21.1 [17.0 to 25.5] | 34.7 [31.8 to NA] — Could not be estimated due to the low number of events
Statistical Analysis 1: Comparison: Placebo + Carboplatin + Paclitaxel -> Placebo vs Veliparib + Carboplatin + Paclitaxel -> Placebo; The secondary efficacy analyses compared investigator-assessed PFS in the Veliparib + Carboplatin + Paclitaxel -> Placebo group (Arm 2) vs. the Placebo + Carboplatin + Paclitaxel -> Placebo group (Arm 1); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.335, Log Rank; Stratified according to residual disease status and disease stage; Hazard Ratio (HR) = 1.215, 95% CI 2-sided [0.821 to 1.799] — Cox proportional hazards model stratified according to the same factors as those used in the log-rank test above

5. Secondary Outcome: Progression-Free Survival (PFS) in the Homologous Recombination Deficiency Cohort (Arm 2 vs Arm 1)
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Veliparib
Number analyzed (Participants) | 207 | 206 | 214
months | 20.5 [17.8 to 22.8] | 18.1 [16.4 to 22.7] | 31.9 [25.8 to 38.0]
Statistical Analysis 1: Comparison: Placebo + Carboplatin + Paclitaxel -> Placebo vs Veliparib + Carboplatin + Paclitaxel -> Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.462, Log Rank; Stratified according to residual disease status and disease stage; Hazard Ratio (HR) = 1.100, 95% CI 2-sided [0.855 to 1.414] — Cox proportional hazards model stratified according to the same factors as those used in the log-rank test above

6. Secondary Outcome: Progression-Free Survival (PFS) in the Intention-to-treat Population (Arm 2 vs Arm 1)
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Veliparib
Number analyzed (Participants) | 375 | 383 | 382
months | 17.3 [15.1 to 19.1] | 15.2 [14.1 to 17.3] | 23.5 [19.3 to 26.3]
Statistical Analysis 1: Comparison: Placebo + Carboplatin + Paclitaxel -> Placebo vs Veliparib + Carboplatin + Paclitaxel -> Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.450, Log Rank; [statistical method as in outcome 3, analysis 1]; Hazard Ratio (HR) = 1.073, 95% CI 2-sided [0.895 to 1.287] — Cox proportional hazards model stratified according to the same factors as those used in the log-rank test above

7. Secondary Outcome: Overall Survival (OS) in the BRCA-deficient Population
Description: OS is defined as the time from the day the participant was randomized to the date of death, and was calculated using Kaplan-Meier methods. All events of death will be included, regardless of whether the event occurs while the participant is still taking study drug, or after discontinuation of study drug. If a participant has not died, then the data will be censored at the date the participant is last known to be alive.
Time Frame: From the time of randomization to the end of the study, up to 98 months
Population: BRCA-Deficient population: All randomized participants with germline and/or tissue deleterious/suspected deleterious BRCA1/2 mutation
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Veliparib
Number analyzed (Participants) | 92 | 98 | 108
months | 89.5 [83.3 to NA] — Could not be estimated due to the low number of events | NA [69.3 to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events
Statistical Analysis 1: Comparison: Placebo + Carboplatin + Paclitaxel -> Placebo vs Veliparib + Carboplatin + Paclitaxel -> Veliparib; Veliparib + Carboplatin + Paclitaxel -> Veliparib (Arm 3) versus Placebo + Carboplatin + Paclitaxel -> Placebo (Arm 1); Test type: Superiority; p = 0.328, Log Rank — Stratified by residual disease (no residual disease after primary surgery versus any residual disease after primary surgery or interval surgery) and stage of disease (stage III versus stage IV); Hazard Ratio (HR) = 0.900, 95% CI 2-sided [0.567 to 1.429] — Cox proportional hazards model stratified according to the same factors as those used in the log-rank test above
Statistical Analysis 2: Comparison: Placebo + Carboplatin + Paclitaxel -> Placebo vs Veliparib + Carboplatin + Paclitaxel -> Placebo; Veliparib + Carboplatin + Paclitaxel -> Placebo (Arm 2) versus Placebo + Carboplatin + Paclitaxel -> Placebo (Arm 1); Test type: Superiority; p = 0.808, Log Rank — [p-value comment as in outcome 7, analysis 1]; Hazard Ratio (HR) = 1.218, 95% CI 2-sided [0.780 to 1.903] — Cox proportional hazards model stratified according to the same factors as those used in the log-rank test above

8. Secondary Outcome: Overall Survival (OS) in the Homologous Recombination Deficiency Population
Description: as for outcome 7
Time Frame: From the time of randomization to the end of the study, up to 98 months
Population: All randomized participants considered BRCA-Deficient and those determined to have HRD tumors based on HRD score
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Veliparib
Number analyzed (Participants) | 207 | 206 | 214
months | 71.5 [59.6 to 87.6] | 74.4 [65.4 to NA] — Could not be estimated due to the low number of events | NA [73.8 to NA] — Could not be estimated due to the low number of events
Statistical Analysis 1: Comparison: Placebo + Carboplatin + Paclitaxel -> Placebo vs Veliparib + Carboplatin + Paclitaxel -> Veliparib; Veliparib + Carboplatin + Paclitaxel -> Veliparib (Arm 3) versus Placebo + Carboplatin + Paclitaxel -> Placebo (Arm 1); Test type: Superiority; p = 0.116, Log Rank — [p-value comment as in outcome 7, analysis 1]; Hazard Ratio (HR) = 0.844, 95% CI 2-sided [0.640 to 1.114] — Cox proportional hazards model stratified according to the same factors as those used in the log-rank test above
Statistical Analysis 2: Comparison: Placebo + Carboplatin + Paclitaxel -> Placebo vs Veliparib + Carboplatin + Paclitaxel -> Placebo; Veliparib + Carboplatin + Paclitaxel -> Placebo (Arm 2) versus Placebo + Carboplatin + Paclitaxel -> Placebo (Arm 1); Test type: Superiority; p = 0.352, Log Rank — [p-value comment as in outcome 7, analysis 1]; Hazard Ratio (HR) = 0.949, 95% CI 2-sided [0.726 to 1.242] — Cox proportional hazards model stratified according to the same factors as those used in the log-rank test above

9. Secondary Outcome: Overall Survival (OS) in the Whole Population
Description: as for outcome 7
Time Frame: From the time of randomization to the end of the study, up to 98 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Veliparib
Number analyzed (Participants) | 375 | 383 | 382
months | 57.8 [52.3 to 63.8] | 58.0 [50.6 to 64.1] | 59.2 [52.1 to 68.2]
Statistical Analysis 1: Comparison: Placebo + Carboplatin + Paclitaxel -> Placebo vs Veliparib + Carboplatin + Paclitaxel -> Veliparib; Veliparib + Carboplatin + Paclitaxel -> Veliparib (Arm 3) versus Placebo + Carboplatin + Paclitaxel -> Placebo (Arm 1); Test type: Superiority; p = 0.283, Log Rank — Stratified by residual disease (none after primary surgery vs any residual disease after primary/interval surgery); disease stage (III vs IV); paclitaxel dosing (Q-weekly vs Q3-weekly); BRCA-Deficient status (Deficient vs wildtype or unknown/missing); Hazard Ratio (HR) = 0.946, 95% CI 2-sided [0.782 to 1.144]
Statistical Analysis 2: Comparison: Placebo + Carboplatin + Paclitaxel -> Placebo vs Veliparib + Carboplatin + Paclitaxel -> Placebo; Veliparib + Carboplatin + Paclitaxel -> Placebo (Arm 2) versus Placebo + Carboplatin + Paclitaxel -> Placebo (Arm 1); Test type: Superiority; p = 0.638, Log Rank — [p-value comment as in outcome 9, analysis 1]; Hazard Ratio (HR) = 1.034, 95% CI 2-sided [0.859 to 1.244] — Cox proportional hazards model stratified according to the same factors as those used in the log-rank test above

10. Secondary Outcome: Change From Baseline in Disease Related Symptom (DRS) Score in the BRCA-mutation Population
Description: The Disease Related Symptom score is a subset of the National Comprehensive Cancer Network Functional Assessment of Cancer Therapy Ovarian Symptom Index-18 (NFOSI-18), which evaluates nine symptoms related to ovarian cancer. The NFOSI-18 DRS score ranges from 0 to 36, with higher scores indicating a lower burden of symptoms and a score of 0 being severely symptomatic. A 3-point difference was defined as clinically meaningful. A positive change from Baseline indicates improvement.
  Change from Baseline was calculated using a used a mixed-model for repeated measures (MMRM) with treatment, stratification factors of residual disease and stage of disease, time point and treatment-by-time point interaction as fixed effect factors, and Baseline DRS score as a covariate.
  DRS was not included in the fixed-sequence testing procedure.
Time Frame: Baseline and Day 1 of Cycles 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, 27, 29, 31, 33, and 35
Population: BRCA-mutation population, participants with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Veliparib
Number analyzed (Participants) | 92 | 98 | 108
score on a scale
  Cycle 3: number analyzed (Participants) | 87 | 84 | 92
  Cycle 3 | 1.8 (0.52) | 0.5 (0.53) | 0.9 (0.51)
  Cycle 5: number analyzed (Participants) | 81 | 80 | 84
  Cycle 5 | 1.7 (0.57) | 0.7 (0.58) | 0.3 (0.56)
  Cycle 7: number analyzed (Participants) | 78 | 84 | 83
  Cycle 7 | 2.6 (0.55) | 1.8 (0.54) | 1.8 (0.54)
  Cycle 9: number analyzed (Participants) | 79 | 80 | 80
  Cycle 9 | 3.3 (0.60) | 3.3 (0.60) | 2.4 (0.59)
  Cycle 11: number analyzed (Participants) | 73 | 81 | 82
  Cycle 11 | 3.2 (0.56) | 3.6 (0.55) | 2.9 (0.54)
  Cycle 13: number analyzed (Participants) | 74 | 80 | 70
  Cycle 13 | 3.6 (0.57) | 3.8 (0.57) | 3.0 (0.57)
  Cycle 15: number analyzed (Participants) | 69 | 63 | 69
  Cycle 15 | 4.3 (0.53) | 4.0 (0.54) | 3.4 (0.52)
  Cycle 17: number analyzed (Participants) | 64 | 66 | 70
  Cycle 17 | 3.8 (0.56) | 4.0 (0.57) | 3.2 (0.55)
  Cycle 19: number analyzed (Participants) | 58 | 53 | 66
  Cycle 19 | 4.0 (0.62) | 4.0 (0.63) | 2.7 (0.59)
  Cycle 21: number analyzed (Participants) | 55 | 56 | 72
  Cycle 21 | 4.6 (0.59) | 3.9 (0.59) | 3.2 (0.55)
  Cycle 23: number analyzed (Participants) | 48 | 47 | 59
  Cycle 23 | 4.2 (0.55) | 4.0 (0.56) | 2.8 (0.52)
  Cycle 25: number analyzed (Participants) | 48 | 45 | 58
  Cycle 25 | 4.0 (0.58) | 5.0 (0.60) | 3.5 (0.55)
  Cycle 27: number analyzed (Participants) | 41 | 42 | 53
  Cycle 27 | 4.5 (0.56) | 4.8 (0.56) | 3.0 (0.52)
  Cycle 29: number analyzed (Participants) | 41 | 39 | 60
  Cycle 29 | 4.0 (0.66) | 5.3 (0.66) | 2.9 (0.59)
  Cycle 31: number analyzed (Participants) | 36 | 36 | 51
  Cycle 31 | 4.8 (0.57) | 4.8 (0.58) | 2.9 (0.52)
  Cycle 33: number analyzed (Participants) | 38 | 38 | 58
  Cycle 33 | 3.9 (0.66) | 5.1 (0.67) | 3.9 (0.59)
  Cycle 35: number analyzed (Participants) | 37 | 37 | 52
  Cycle 35 | 4.5 (0.61) | 5.0 (0.62) | 3.2 (0.56)

11. Secondary Outcome: Change From Baseline in Disease Related Symptom (DRS) Score in the HRD Population
Description: as for outcome 10
Time Frame: Baseline and Day 1 of Cycles 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, 27, 29, 31, 33, and 35
Population: HRD population, participants with available data at each time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Veliparib
Number analyzed (Participants) | 207 | 206 | 214
score on a scale
  Cycle 3: number analyzed (Participants) | 187 | 179 | 186
  Cycle 3 | 1.5 (0.35) | 0.5 (0.36) | 0.9 (0.35)
  Cycle 5: number analyzed (Participants) | 178 | 169 | 172
  Cycle 5 | 1.7 (0.37) | 1.1 (0.37) | 0.8 (0.37)
  Cycle 7: number analyzed (Participants) | 172 | 168 | 170
  Cycle 7 | 2.4 (0.35) | 1.8 (0.36) | 2.2 (0.35)
  Cycle 9: number analyzed (Participants) | 173 | 165 | 165
  Cycle 9 | 3.3 (0.37) | 3.6 (0.38) | 2.3 (0.38)
  Cycle 11: number analyzed (Participants) | 162 | 161 | 159
  Cycle 11 | 3.5 (0.36) | 3.5 (0.36) | 2.7 (0.36)
  Cycle 13: number analyzed (Participants) | 160 | 159 | 134
  Cycle 13 | 3.6 (0.37) | 3.8 (0.38) | 2.7 (0.39)
  Cycle 15: number analyzed (Participants) | 149 | 138 | 130
  Cycle 15 | 4.2 (0.35) | 3.9 (0.36) | 3.3 (0.37)
  Cycle 17: number analyzed (Participants) | 139 | 129 | 124
  Cycle 17 | 3.9 (0.39) | 3.4 (0.40) | 3.0 (0.40)
  Cycle 19: number analyzed (Participants) | 120 | 107 | 119
  Cycle 19 | 4.2 (0.40) | 3.7 (0.42) | 2.7 (0.41)
  Cycle 21: number analyzed (Participants) | 115 | 110 | 118
  Cycle 21 | 4.6 (0.40) | 3.6 (0.41) | 3.0 (0.40)
  Cycle 23: number analyzed (Participants) | 105 | 95 | 103
  Cycle 23 | 4.1 (0.38) | 3.6 (0.39) | 3.1 (0.38)
  Cycle 25: number analyzed (Participants) | 99 | 86 | 96
  Cycle 25 | 4.1 (0.40) | 4.4 (0.41) | 3.5 (0.40)
  Cycle 27: number analyzed (Participants) | 88 | 81 | 87
  Cycle 27 | 4.4 (0.39) | 4.4 (0.40) | 3.0 (0.38)
  Cycle 29: number analyzed (Participants) | 86 | 76 | 96
  Cycle 29 | 4.2 (0.43) | 4.7 (0.44) | 3.2 (0.41)
  Cycle 31: number analyzed (Participants) | 78 | 73 | 82
  Cycle 31 | 3.9 (0.41) | 4.3 (0.42) | 3.3 (0.40)
  Cycle 33: number analyzed (Participants) | 73 | 74 | 89
  Cycle 33 | 4.2 (0.45) | 4.7 (0.45) | 3.9 (0.42)
  Cycle 35: number analyzed (Participants) | 68 | 69 | 78
  Cycle 35 | 4.1 (0.44) | 4.6 (0.45) | 3.4 (0.43)

12. Secondary Outcome: Change From Baseline in Disease Related Symptom (DRS) Score in the Whole Population
Description: The Disease Related Symptom score is a subset of the National Comprehensive Cancer Network Functional Assessment of Cancer Therapy Ovarian Symptom Index-18 (NFOSI-18), which evaluates nine symptoms related to ovarian cancer. The NFOSI-18 DRS score ranges from 0 to 36, with higher scores indicating a lower burden of symptoms and a score of 0 being severely symptomatic. A 3-point difference was defined as clinically meaningful. A positive change from Baseline indicates improvement.
  Change from Baseline was calculated using a used a mixed-model for repeated measures (MMRM) with treatment, stratification factors of residual disease, stage of disease, choice of paclitaxel dosing regimen and BRCA-deficient status, time point and treatment-by-time point interaction as fixed effect factors, and Baseline DRS score as a covariate.
  DRS was not included in the fixed-sequence testing procedure.
Time Frame: Baseline and Day 1 of Cycles 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, 27, 29, 31, 33, and 35
Population: All randomized participants with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Veliparib
Number analyzed (Participants) | 375 | 383 | 382
score on a scale
  Cycle 3: number analyzed (Participants) | 333 | 332 | 320
  Cycle 3 | 1.5 (0.28) | 0.4 (0.28) | 0.9 (0.28)
  Cycle 5: number analyzed (Participants) | 310 | 312 | 301
  Cycle 5 | 1.6 (0.29) | 0.9 (0.29) | 0.8 (0.29)
  Cycle 7: number analyzed (Participants) | 300 | 301 | 287
  Cycle 7 | 2.3 (0.29) | 1.8 (0.29) | 2.1 (0.29)
  Cycle 9: number analyzed (Participants) | 291 | 290 | 277
  Cycle 9 | 3.3 (0.29) | 3.8 (0.29) | 2.4 (0.29)
  Cycle 11: number analyzed (Participants) | 270 | 267 | 249
  Cycle 11 | 3.5 (0.29) | 4.0 (0.28) | 3.0 (0.29)
  Cycle 13: number analyzed (Participants) | 254 | 254 | 225
  Cycle 13 | 3.8 (0.30) | 4.0 (0.30) | 3.2 (0.30)
  Cycle 15: number analyzed (Participants) | 224 | 226 | 207
  Cycle 15 | 4.2 (0.30) | 3.8 (0.30) | 3.3 (0.30)
  Cycle 17: number analyzed (Participants) | 204 | 203 | 202
  Cycle 17 | 4.1 (0.32) | 3.7 (0.32) | 3.4 (0.32)
  Cycle 19: number analyzed (Participants) | 177 | 171 | 178
  Cycle 19 | 4.4 (0.32) | 4.0 (0.32) | 3.1 (0.32)
  Cycle 21: number analyzed (Participants) | 170 | 160 | 174
  Cycle 21 | 4.3 (0.34) | 3.6 (0.34) | 3.3 (0.33)
  Cycle 23: number analyzed (Participants) | 151 | 139 | 154
  Cycle 23 | 4.0 (0.33) | 3.9 (0.33) | 3.3 (0.32)
  Cycle 25: number analyzed (Participants) | 145 | 127 | 145
  Cycle 25 | 4.0 (0.34) | 4.1 (0.35) | 3.5 (0.33)
  Cycle 27: number analyzed (Participants) | 129 | 120 | 130
  Cycle 27 | 4.4 (0.33) | 4.2 (0.34) | 3.5 (0.32)
  Cycle 29: number analyzed (Participants) | 123 | 114 | 136
  Cycle 29 | 4.4 (0.34) | 4.4 (0.35) | 3.4 (0.33)
  Cycle 31: number analyzed (Participants) | 112 | 109 | 120
  Cycle 31 | 4.0 (0.36) | 4.2 (0.37) | 3.3 (0.35)
  Cycle 33: number analyzed (Participants) | 106 | 105 | 123
  Cycle 33 | 4.1 (0.38) | 4.4 (0.38) | 3.7 (0.36)
  Cycle 35: number analyzed (Participants) | 99 | 100 | 111
  Cycle 35 | 4.4 (0.37) | 4.2 (0.37) | 3.7 (0.35)

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse events were collected from the time informed consent was signed through the end of the study. Median time on follow-up was 81.7 months for the Placebo + Carboplatin + Paclitaxel -> Placebo group, 81.2 months for the Veliparib + Carboplatin + Paclitaxel -> Placebo group, and 81.1 months for the Veliparib + Carboplatin + Paclitaxel -> Veliparib group.
Groups:
- Veliparib + Carboplatin + Paclitaxel -> Veliparib: Participants received 150 mg veliparib orally twice a day in combination with carboplatin given at an AUC of 6 mg/mL/min every 3 weeks, and paclitaxel 175 mg/m² of BSA administered every 3 weeks, or 80 mg/m² administered weekly, for six 21-day cycles.
  Participants who completed chemotherapy without disease progression received single-agent\ veliparib at a dose of 300 mg twice daily for 2 weeks (transition period) and then 400 mg veliparib twice daily if the dose in the transition period was not associated with limiting side effects for an additional thirty 21-day cycles of maintenance therapy.
Arm/Group | Placebo + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Placebo | Veliparib + Carboplatin + Paclitaxel -> Veliparib
All-Cause Mortality (participants affected / at risk) | 228/375 | 234/383 | 209/382
Serious Adverse Events (participants affected / at risk) | 143/375 | 130/383 | 146/382
Other Adverse Events (participants affected / at risk) | 369/375 | 375/383 | 376/382
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Carboplatin + Paclitaxel -> Placebo (N=375) | Veliparib + Carboplatin + Paclitaxel -> Placebo (N=383) | Veliparib + Carboplatin + Paclitaxel -> Veliparib (N=382)
ANAEMIA (Blood and lymphatic system disorders) | 4 (4) | 13 (14) | 14 (18)
APLASTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
BONE MARROW FAILURE (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 9 (10) | 19 (20) | 15 (17)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 6 (9) | 16 (22) | 12 (16)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 (3) | 9 (12) | 10 (20)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 3 (3) | 1 (2) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
PALPITATIONS (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
STRESS CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
VISION BLURRED (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL ADHESIONS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
ABDOMINAL INCARCERATED HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 (5) | 9 (10) | 9 (10)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ASCITES (Gastrointestinal disorders) | 7 (9) | 3 (3) | 2 (2)
COLITIS (Gastrointestinal disorders) | 1 (2) | 3 (3) | 1 (1)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 3 (3) | 5 (5) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 4 (5) | 2 (2)
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ENTEROCOLITIS (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
EPIPLOIC APPENDAGITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTRIC VOLVULUS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
HAEMOPERITONEUM (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
HIATUS HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ILEAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
ILEUS (Gastrointestinal disorders) | 2 (2) | 7 (7) | 3 (4)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 (4) | 1 (1) | 6 (7)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
INTESTINAL PSEUDO-OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
INTRA-ABDOMINAL FLUID COLLECTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 2 (3) | 1 (1)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
MECHANICAL ILEUS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 4 (5) | 11 (11) | 13 (16)
OESOPHAGITIS ULCERATIVE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PNEUMOPERITONEUM (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 19 (22) | 13 (17) | 11 (14)
SMALL INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
SPIGELIAN HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 5 (5) | 10 (10) | 12 (16)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 1 (1)
CHEST DISCOMFORT (General disorders) | 0 (0) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0)
CHILLS (General disorders) | 0 (0) | 0 (0) | 2 (2)
DISEASE PROGRESSION (General disorders) | 0 (0) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 2 (3)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 0 (0) | 1 (1)
HERNIA (General disorders) | 1 (1) | 0 (0) | 0 (0)
IMPLANT SITE EXTRAVASATION (General disorders) | 0 (0) | 0 (0) | 1 (1)
INCARCERATED HERNIA (General disorders) | 1 (1) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 4 (4)
PAIN (General disorders) | 1 (1) | 0 (0) | 1 (1)
PELVIC MASS (General disorders) | 0 (0) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 6 (6) | 3 (3) | 9 (9)
BILE DUCT STONE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
ANAPHYLACTIC REACTION (Immune system disorders) | 1 (1) | 1 (1) | 1 (1)
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 2 (2) | 2 (2)
ABDOMINAL ABSCESS (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
ATYPICAL MYCOBACTERIAL INFECTION (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
BACTERAEMIA (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
BACTEROIDES BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
CATHETER SITE INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 3 (4) | 2 (2) | 1 (1)
COLONIC ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CYSTITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
DEVICE RELATED INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
EMPYEMA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ENDOCARDITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ENTEROBACTER INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ENTEROCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
ERYSIPELAS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ESCHERICHIA INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
GROIN ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
IMPLANT SITE INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
INFECTED LYMPHOCELE (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
INFLUENZA (Infections and infestations) | 0 (0) | 3 (3) | 3 (3)
INTERVERTEBRAL DISCITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
KIDNEY INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
LARGE INTESTINE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
LYMPHANGITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
MENINGITIS CRYPTOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
NAIL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
NEUTROPENIC SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OPHTHALMIC HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
OSTEOMYELITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PELVIC ABSCESS (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
PELVIC INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PERIORBITAL CELLULITIS (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
PERITONEAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
PERITONITIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PHLEBITIS INFECTIVE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 6 (7) | 5 (5) | 4 (5)
PNEUMONIA ASPIRATION (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
POST PROCEDURAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
POSTOPERATIVE ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 (1) | 2 (2) | 1 (2)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 7 (7) | 3 (3) | 5 (6)
SEPTIC EMBOLUS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 5 (6) | 3 (3) | 4 (5)
SPONTANEOUS BACTERIAL PERITONITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SUBDIAPHRAGMATIC ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SYSTEMIC CANDIDA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 4 (5) | 6 (6) | 7 (7)
UROSEPSIS (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
WOUND INFECTION (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
ACETABULUM FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
CONCUSSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 7 (7) | 0 (0) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
FRACTURED SACRUM (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL STOMA COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
HEAT ILLNESS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
INTESTINAL ANASTOMOSIS COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
SKELETAL INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
VAGINAL CUFF DEHISCENCE (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
WOUND DECOMPOSITION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
SOLUBLE FIBRIN MONOMER COMPLEX INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 6 (6) | 0 (0) | 6 (6)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 6 (7)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (3)
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (14) | 11 (13) | 5 (6)
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2)
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
CEREBELLAR INFARCTION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
CEREBRAL ARTERY EMBOLISM (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
CEREBRAL VENOUS SINUS THROMBOSIS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERSOMNIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
MIGRAINE WITH AURA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
NEURALGIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 6 (6) | 1 (1) | 6 (6)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
DEVICE BREAKAGE (Product Issues) | 1 (1) | 0 (0) | 0 (0)
DEVICE DISLOCATION (Product Issues) | 0 (0) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 (2) | 1 (1) | 2 (2)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
RENAL INFARCT (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
RENAL VEIN THROMBOSIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
URETEROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
FEMALE GENITAL TRACT FISTULA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
DYSPNOEA AT REST (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (7) | 0 (0)
PNEUMONITIS ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
PNEUMOTHORAX SPONTANEOUS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 10 (11) | 12 (13)
PULMONARY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2) | 2 (2) | 4 (4)
EMBOLISM (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 2 (2) | 1 (1)
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 2 (2) | 0 (0) | 2 (2)
LYMPHOCELE (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
PHLEBITIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
SUBCLAVIAN VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
THROMBOPHLEBITIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
VENOUS THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Carboplatin + Paclitaxel -> Placebo (N=375) | Veliparib + Carboplatin + Paclitaxel -> Placebo (N=383) | Veliparib + Carboplatin + Paclitaxel -> Veliparib (N=382)
ANAEMIA (Blood and lymphatic system disorders) | 191 (514) | 232 (603) | 226 (672)
LEUKOPENIA (Blood and lymphatic system disorders) | 89 (223) | 87 (261) | 114 (333)
LYMPHOPENIA (Blood and lymphatic system disorders) | 15 (28) | 15 (20) | 26 (57)
NEUTROPENIA (Blood and lymphatic system disorders) | 247 (673) | 266 (881) | 273 (848)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 119 (266) | 216 (630) | 209 (735)
VISION BLURRED (Eye disorders) | 32 (33) | 19 (22) | 27 (27)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 45 (55) | 48 (54) | 34 (39)
ABDOMINAL PAIN (Gastrointestinal disorders) | 114 (163) | 105 (143) | 118 (162)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 29 (38) | 18 (24) | 29 (37)
CONSTIPATION (Gastrointestinal disorders) | 157 (203) | 177 (241) | 165 (228)
DIARRHOEA (Gastrointestinal disorders) | 149 (248) | 137 (228) | 164 (255)
DRY MOUTH (Gastrointestinal disorders) | 19 (20) | 10 (12) | 22 (23)
DYSPEPSIA (Gastrointestinal disorders) | 41 (53) | 45 (55) | 36 (42)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 22 (23) | 28 (30) | 34 (46)
NAUSEA (Gastrointestinal disorders) | 246 (425) | 259 (433) | 289 (578)
STOMATITIS (Gastrointestinal disorders) | 52 (67) | 47 (52) | 59 (67)
VOMITING (Gastrointestinal disorders) | 128 (211) | 123 (170) | 174 (309)
ASTHENIA (General disorders) | 28 (58) | 36 (56) | 41 (64)
FATIGUE (General disorders) | 221 (353) | 235 (407) | 257 (456)
MALAISE (General disorders) | 21 (34) | 22 (31) | 31 (37)
MUCOSAL INFLAMMATION (General disorders) | 19 (21) | 16 (18) | 18 (21)
OEDEMA PERIPHERAL (General disorders) | 73 (84) | 58 (62) | 56 (77)
PAIN (General disorders) | 22 (25) | 22 (31) | 21 (23)
PYREXIA (General disorders) | 25 (28) | 33 (38) | 23 (30)
DRUG HYPERSENSITIVITY (Immune system disorders) | 63 (84) | 48 (63) | 51 (56)
NASOPHARYNGITIS (Infections and infestations) | 21 (26) | 19 (22) | 26 (32)
SINUSITIS (Infections and infestations) | 18 (27) | 18 (20) | 21 (22)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 43 (52) | 28 (36) | 34 (44)
URINARY TRACT INFECTION (Infections and infestations) | 67 (104) | 64 (91) | 70 (91)
CONTUSION (Injury, poisoning and procedural complications) | 13 (13) | 17 (21) | 20 (28)
FALL (Injury, poisoning and procedural complications) | 19 (20) | 15 (16) | 18 (23)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 37 (46) | 18 (19) | 25 (25)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 41 (64) | 31 (55) | 40 (52)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 31 (46) | 22 (41) | 31 (35)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 19 (26) | 10 (13) | 16 (21)
WEIGHT DECREASED (Investigations) | 32 (45) | 41 (52) | 54 (71)
WEIGHT INCREASED (Investigations) | 35 (49) | 26 (34) | 36 (52)
DECREASED APPETITE (Metabolism and nutrition disorders) | 85 (101) | 82 (106) | 110 (143)
DEHYDRATION (Metabolism and nutrition disorders) | 20 (21) | 32 (48) | 30 (37)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 18 (35) | 18 (26) | 27 (50)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 19 (31) | 12 (17) | 16 (31)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 69 (107) | 68 (113) | 59 (94)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 98 (199) | 96 (142) | 85 (143)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 25 (33) | 21 (24) | 25 (35)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 21 (31) | 14 (18) | 11 (14)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 136 (217) | 112 (152) | 114 (166)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 66 (87) | 66 (75) | 67 (88)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 27 (46) | 25 (36) | 33 (37)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 23 (28) | 24 (34) | 23 (33)
MYALGIA (Musculoskeletal and connective tissue disorders) | 75 (106) | 59 (80) | 71 (96)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 55 (70) | 46 (56) | 51 (64)
DIZZINESS (Nervous system disorders) | 90 (121) | 83 (105) | 100 (126)
DYSGEUSIA (Nervous system disorders) | 57 (70) | 47 (54) | 73 (80)
HEADACHE (Nervous system disorders) | 97 (136) | 90 (124) | 98 (143)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 256 (415) | 235 (346) | 242 (373)
TREMOR (Nervous system disorders) | 9 (11) | 6 (6) | 23 (26)
ANXIETY (Psychiatric disorders) | 58 (72) | 61 (74) | 59 (70)
DEPRESSION (Psychiatric disorders) | 39 (46) | 46 (58) | 34 (43)
INSOMNIA (Psychiatric disorders) | 89 (105) | 120 (141) | 109 (134)
DYSURIA (Renal and urinary disorders) | 22 (24) | 17 (18) | 16 (17)
COUGH (Respiratory, thoracic and mediastinal disorders) | 58 (70) | 57 (63) | 59 (70)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 76 (106) | 91 (112) | 84 (111)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 59 (70) | 61 (66) | 56 (61)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 26 (29) | 6 (6) | 18 (22)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 39 (46) | 24 (27) | 27 (33)
ALOPECIA (Skin and subcutaneous tissue disorders) | 214 (271) | 216 (271) | 197 (256)
NAIL DISCOLOURATION (Skin and subcutaneous tissue disorders) | 21 (21) | 10 (10) | 9 (9)
PRURITUS (Skin and subcutaneous tissue disorders) | 40 (49) | 35 (41) | 28 (33)
RASH (Skin and subcutaneous tissue disorders) | 56 (68) | 54 (64) | 48 (53)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 30 (35) | 11 (15) | 22 (31)
HOT FLUSH (Vascular disorders) | 49 (53) | 44 (48) | 43 (50)
HYPERTENSION (Vascular disorders) | 38 (66) | 38 (60) | 32 (60)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT02470585/Prot_002.pdf
  • Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/85/NCT02470585/SAP_001.pdf